CLINICAL TRIAL: NCT04368819
Title: A Single-center, Randomized, Double-blind, Placebo-controlled Study of the Efficacy and Safety of Allopurinol in Improving Ischemic Symptoms in Patients With Refractory Angina.
Brief Title: Allopurinol in Patients With Refractory Angina to Improve Ischemic Symptoms
Acronym: ARAMIS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health, Brazil (Other Government)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Luis Henrique W Gowdak, MD, PhD, Clinical Scientist, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SDC 4781/18/132; 2018/22588-3 (Other Grant/Funding Number: Fundação de Amparo à Pesquisa do Estado de São Paulo)
Record Dates: First submitted 2020-04-23; First posted 2020-04-30 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Refractory Angina
Keywords: angina; coronary artery disease; myocardial ischemia; treatment; allopurinol; cardiopulmonary exercising test; oxidative stress; stress echocardiogram
MeSH Terms: conditions — Angina Pectoris; Coronary Artery Disease; Myocardial Ischemia | interventions — Allopurinol

STUDY DESIGN:
Intervention Model Description: Patients will randomly be assigned to receive either placebo or allopurinol 300mg once daily for four weeks, up titrate to 600mg for another 12 weeks for a total of 16 weeks of treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo pills will be manufactured to be indistinguishable from the active treatment and dispensed by a registered pharmacist (who also will be blind to the intervention assigned to each individual participant) from our center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allopurinol (Active Comparator): Allopurinol 300mg P.O. once daily for four weeks followed by allopurinol 300mg P.O. twice daily for 12 weeks.
  Interventions: Drug: Allopurinol 300 MG
- Placebo (Placebo Comparator): Placebo pills indistinguishable from the active comparator given P.O. once daily for four weeks, followed by twice daily for 12 weeks.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Allopurinol 300 MG — Allopurinol 300mg once daily for four weeks followed by allopurinol 300mg twice daily for 12 weeks
  Other Names: Zyloric
  Arms: Allopurinol
Drug: Placebo oral tablet — Placebo 300mg once daily for four weeks followed by allopurinol 300mg twice daily for 12 weeks
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Despite numerous advances in medical treatment and revascularization procedures for the treatment of patients with stable angina, debilitating symptoms that are unresponsive to conventional therapy may occur in patients unsuitable for revascularization, a condition known as refractory angina. Allopurinol, a methylxanthine oxidase inhibitor, is widely used in the treatment of gout and asymptomatic hyperuricemia. On the other hand, the anti-ischemic effects of allopurinol have been the subject of increasing interest. Therefore, the investigators will study the safety and efficacy of allopurinol in alleviating ischemic symptoms in patients with refractory angina already on optimal medical therapy.

DETAILED DESCRIPTION:
One of the most common clinical presentations associated with coronary artery disease (CAD) is stable angina, which can be translated clinically into chest discomfort (or equivalent) evoked by different levels of physical activity depending on the extent of the disease. In the United States, it is estimated that 16.5 million individuals over 20 years of age have chronic ischemic heart disease, of which 3.4 million live with the diagnosis of angina pectoris. Refractory angina is a clinical condition characterized by the presence of debilitating symptoms secondary to CAD lasting more than three months in which the symptoms are attributed to objectively documented ischemia and not controlled with the combination of conventional antianginal agents and myocardial revascularization procedures. The estimated annual incidence of patients with refractory angina is between 50,000 and 200,000 new cases in the United States.

Allopurinol, a methylxanthine oxidase inhibitor, is widely used in the treatment of gout and asymptomatic hyperuricemia. The therapeutic potential of allopurinol in patients with cardiovascular disease has been the subject of increasing interest. In patients with CAD, the first study tested the role of allopurinol in improving exercise tolerance in 65 patients with stable angina documented by angiography and positive stress test for myocardial ischemia. After only six weeks of treatment, patients who received allopurinol showed a statistically significant increase in ergometry parameters, including time for ST-segment depression, total exercise time, and time until the onset of angina. There were no reports of adverse events. Considerable decrease in inflammatory markers and oxidative stress indicators has been demonstrated in patients with acute myocardial infarction receiving allopurinol versus placebo with a significant reduction in the risk of cardiovascular events in 2 years (10% vs. 30%, respectively). Therefore, the investigators will test the hypothesis that the use of allopurinol increases exercise tolerance and reduces angina attacks compared to placebo after 16 weeks of follow-up in patients with refractory angina.

Patients will be randomly selected to receive a placebo or allopurinol (600mg od) for 16 weeks. At baseline and after 16 weeks of treatment, exercise tolerance will be assessed through the cardiopulmonary exercising test, and myocardial ischemia will be determined using an exercise echocardiogram protocol. Biomarkers of oxidative stress will be measured in the blood and urine; endothelial-dependent vasodilation will be assessed using the reactive hyperemia protocol at the brachial artery.

For the sample size calculation, the investigators chose the primary outcome as "total exercise time (TTE) after intervention" based on the study by Noman et al. (Lancet 2010;375:2161-7). Thus, assuming that μ1 (allopurinol) = 396sec, μ2 (placebo) = 319sec and σ = 63sec, the investigators concluded that to be able to detect a difference between groups with 95% confidence (1-alfa) and 90% power (1-beta), 17 patients are needed in each study group. If the investigators consider a screen failure rate at 20%, a total of 40 patients will be needed, randomized 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stable angina in functional class (CCS) ≥ 2 for at least three months in patients taking maximally tolerated doses of at least three classes of antianginal agents
* Documentation of myocardial ischemia by any provocative functional test (exercise test, stress echocardiogram, myocardial perfusion scintigraphy or cardiac resonance)
* Signature of the Informed Consent Form

Exclusion Criteria:

* Left ventricular dysfunction defined by LVEF < 30% on transthoracic echocardiogram
* Significant concomitant valve disease
* Chronic renal failure stage 4 or 5 (GFR < 30mL/min/1.73m2 calculated by the MDRD equation
* Significant liver dysfunction (Child-Pugh class C) or MELD value ≥ 15 calculated from creatinine, total bilirubin, and INR values
* Current use of warfarin
* Prior use of allopurinol within three months of randomization
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-03 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Increase in total exercise time (seconds) assessed by CPET | 16 weeks
  Total exercise duration during a maximal, symptom-limited cardiopulmonary exercise testing

SECONDARY OUTCOMES:
Number of angina attacks per week | 16 weeks
  Frequency of patient-reported daily diary of angina
Short-acting nitrates intake per week | 16 weeks
  Frequency of patient-reported short-acting nitrates intake for symptom-relief
Relative decrease in stress-induced myocardial ischemia during exercise echocardiogram | 16 weeks
  % of change in myocardial ischemia burden assessed during exercise echocardiogram stress test compared to baseline
Relative change in the levels of oxidative stress biomarkers | 16 weeks
  % of change in the level of biomarkers of stress oxidative (nitrotyrosine, malondialdehyde and of reduced glutathione) compared to baseline
Relative change in endothelium-dependent vasodilation during reactive hyperemia in the forearm | 16 weeks
  % of improvement in endothelium-dependent vasodilation assessed during reactive hyperemia (brachial artery) compared to baseline

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 16 weeks
  All AE will be recorded during the 16 week period of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Luis Henrique W Gowdak, MD, PhD, Principal Investigator — Heart Institute (InCor-HCFMUSP)
Locations (1):
- Heart Institute, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
We must abide by the local regulations.

REFERENCES:
- [Background] Noman A, Ang DS, Ogston S, Lang CC, Struthers AD. Effect of high-dose allopurinol on exercise in patients with chronic stable angina: a randomised, placebo controlled crossover trial. Lancet. 2010 Jun 19;375(9732):2161-7. doi: 10.1016/S0140-6736(10)60391-1. Epub 2010 Jun 9. PMID 20542554